CLINICAL TRIAL: NCT02199912
Title: ANC2 Pilot Study Study of the Relationship Between Clinical and Paraclinical Markers During Situations of Cachexia and Pre-cachexia in Patients Over 70 Years With Colorectal Surgery
Brief Title: Study of the Relationship Between Clinical and Paraclinical Markers During Situations of Cachexia and Pre-cachexia in Patients Over 70 Years With Colorectal Surgery
Acronym: ANC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012.752; 2012-A01017-36 (Registry Identifier: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2014-06-26; First posted 2014-07-25 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Tumor
Keywords: cachexia; nutrition; cancer; colorectal tumor
MeSH Terms: conditions — Colorectal Neoplasms; Cachexia; Neoplasms | interventions — Blood Specimen Collection; Calorimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with colorectal surgery (Experimental)
  Interventions: Procedure: Biopsy of adipose and muscular tissue; Other: Blood sampling; Other: Calorimetry; Other: Impedance measure; Other: Evaluation of nutritional status; Other: Evaluation of physical performance; Other: Evaluation of muscular strength; Other: Evaluation of emotional status; Other: Evaluation of functional status

INTERVENTIONS:
Procedure: Biopsy of adipose and muscular tissue
Other: Blood sampling
Other: Calorimetry
Other: Impedance measure — Evaluation of physical composition (non-invasive method)
Other: Evaluation of nutritional status — Nutritional status will be assessed by using the "Mini Nutritional Assessment" (MNA) questionnaire and a scale that evaluates anorexia
Other: Evaluation of physical performance — This will be assessed by using a "tiredness scale" named "Echelle Visuelle Analogique" (EVA) in french
Other: Evaluation of muscular strength — Muscular strength will be assessed thanks to the Handgrip Strength Test and the Short Physical Performance Battery (SPPB)
Other: Evaluation of emotional status — The emotional status wil be assessed thanks to the Yesavage Geriatric Depression Scale (GDS)
Other: Evaluation of functional status — The functional status will be assessed by using the Activity of Daily Life (ADL) questionnaire and the Instrumental Activities of Daily Living (IADL) Questionnaire

SUMMARY:
Cachexia associated with cancer is a grave and most of the time irreversible common situation. It seems independent from the size of the tumor or from its metastatic character. The consequences for the management of the patient are major and exceed widely the frame of the nutrition.

Undernutrition of patients with cancer is described by a decrease of the energy contributions and a loss of muscular and fat mass, leading to a progressive functional deficiency which can go to the cachectic state.

Actually, clinical criteria are proposed allowing to characterize the state of pre-cachexia but it remain too indistinct to allow an early and efficient screening and set up effective measures of prevention of the cachexia, to avoid the loss of muscular tissue and the cast iron of the energy reserves.

It is necessary to have clinical and biological markers with diagnostic aim and forecasts during the situations precedents the appearance of cachexia.

The present study will allow calibrating a longitudinal study, which could confirm the value of measures made for the diagnosis of pre-cachexia.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 70 years
* Colorectal tumor resection with/without synchronous metastases

Exclusion Criteria:

* Emergency resection of colorectal tumor
* Unresectable colorectal tumor with/without synchronous metastases

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
biological and radiological markers | During perioperative period (from date of consent until discharge from the hospital, up to 30 postoperative days)
  Validated criteria of cachexia, pre-cachexia and sarcopenia are applied. Systematic preoperative measures (TNFα, leptin, ghrelin) and CT scanning of the abdomen/pelvis are performed for all patient enrolled.

SECONDARY OUTCOMES:
activity of the ATGL | During perioperative period (From date of consent until discharge from the hospital, up to 30 postoperative days)
  The activity of ATGL is determined by liquid scintillation counting.
Body composition | During perioperative period (from date of consent until discharge from the hospital, up to 30 postoperative days)
  Body composition is evaluated utilizing computerized tomography(CT) images (at the third lumbar vertebral level). A muscle index is also calculated by normalizing muscle areas for height.
metabolic phenotype | During perioperative period (From date of consent until discharge from the hospital, up to 30 postoperative days)
  metabolic phenotype is determinated by indirect calorimetry.
loss of fat body mass and/or lean body mass | During perioperative period (From date of consent until discharge from the hospital, up to 30 postoperative days)
  Lean body mass and components (intracellular water and extracellular water as well as body cell mass) were calculated by tetrapolar bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Sud - Service de Médecine Gériatrique, Pierre-Bénite, France